CLINICAL TRIAL: NCT02247986
Title: Investigating the Impact of Methylphenidate on Neural Response in Disruptive Behavioral Disorder
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 140193; 14-M-0193
Record Dates: First submitted 2014-09-20; First posted 2014-09-25 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2015-05-18

CONDITIONS: Conduct Disorder; Attention Defict Hyperactivity Disorder
Keywords: Conduct Disorder; Methylphenidate; Disruptive Behavior Disorders
MeSH Terms: conditions — Conduct Disorder; Attention Deficit and Disruptive Behavior Disorders | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Methylphenidate Hydrochloride — Bold signal changes by methylphenidate on DBD

SUMMARY:
Background:

- Disruptive behavior is a common problem for children and adolescents. It can be treated with some success with stimulant medicine. Researchers want to learn more about how this works.

Objective:

- To learn how the brain changes when taking the medicine methylphenidate for behavior problems.

Eligibility:

* Children ages 10 17 with conduct disorder and/or attention deficit disorder.
* Healthy volunteers the same age.

Design:

* Participants will be screened under a separate protocol.
* Participants will have two 3-hour sessions at the clinic. Girls who are menstruating will have a pregnancy test before their scans.
* Visit 1: All participants will:
* Perform simple tests on a computer.
* Fill out a questionnaire along with their parent or guardian.
* Have an MRI scan. A magnetic field and radio waves take pictures of the brain. Participants will lie on a table that slides into a metal cylinder. A coil will be placed over their head. They will be in the scanner for 60 minutes, lying still or performing a simple task. They will practice the task before the scan. A computer screen will show them task information during the scan. The scanner makes loud knocking sounds. Participants will get earplugs. Their parent or guardian can stay with them during the scan.
* Only participants with behavior disorders will:
* Take a pill of the study medicine or placebo.
* Be monitored for any side effects.
* Visit 2 is a repeat of Visit 1, except participants who got a pill in Visit 1 will get the other pill in Visit 2. For healthy volunteers, the 2 visits are exactly the same.

DETAILED DESCRIPTION:
OBJECTIVE:

To determine the impact, as indexed by BOLD response, of the administration of dopaminergic agonist (methylphenidate) on the pathophysiology of CD/ODD.

STUDY POPULATION:

Youth with CD/ODD and typically developing (TD) youth.

DESIGN:

The study will involve a 2 session design (methylphenidate [MPH] vs. placebo). Patients with CD/ODD will participate in both sessions. TD youth will be tested for 2 sessions (no medication) to provide an index of typical task response. Activity within regions of interest identified from the TD youth will be used to determine whether MPH reduces differences in BOLD response in CD/ODD relative to TD youth. ICU scores and current ADHD symptomatology will be used as covariates to determine whether these variables moderate the putative increase in BOLD response in target regions in the patients with CD.

OUTCOME MEASURES:

Principle dependent measures will be BOLD responses as measured through core tasks.

ELIGIBILITY:
* INCLUSION CRITERIA

Youth with CD

1. 10-17 years of age.
2. A current diagnosis of CD as determined by the Kiddie-SADS, lifetime version.

   * Youth in the CD+comorbid ADHD group will also meet diagnostic criteria for ADHD.
   * Youth in the CD without comorbid ADHD group will specifically not meet diagnostic criteria for ADHD.
3. Youth with CD shouldmust be na(SqrRoot) ve to psychoactive medication (such as: methylphenidate and amphetamine).

TD youth

1. 10-17 years of age.
2. No current psychiatric diagnosis, as determined by the Kiddie-SADS, lifetime version.

EXCLUSION CRITERIA

Exclusion criteria for youth with CD (with or without ADHD)

1. Comorbid psychotic, major mood, tic, pervasive developmental, and substance abuse disorders.
2. Presence of comorbid ADHD is exclusory for the group of patients with CD without ADHD
3. History of known structural cardiac abnormalities, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, or other serious cardiac problems
4. Current weight less than 25kg or over 90kg

Exclusion criteria for all participants (CD with ADHD, CD without ADHD and TD)

1. History of serious CNS disease disorder (examples aresuch as: history of seizure, epilepsy, brain tumor, brain hemorrhage, and major CNS infection such as meningitis or encephalitis)
2. Previous history of known structural cardiac abnormalities, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, or other serious cardiac problems
3. Current use of any psychiatric medications and centrally acting medications (such as stimulants, non-stimulant ADHD medications, antidepressants, anxiolytics, antipsychotics and anti-epilepsy medications), and past history of use of psychoactive medication (such as methylphenidate and amphetamine)
4. A positive urine pregnancy test
5. A Positive urine toxicology, History/current diagnosis of substance abuse/dependence
6. Suicidal or homicidal ideation within the past 6 months.
7. Wechsler Abbreviated Scale of Intelligence (WASI) (D. Wechsler, 1999) scores <70
8. Metal in body (i.e., hearing aid, cardiac pacemaker, bone plates, etc), claustrophobia, or any other condition that would preclude fMRI scanning.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-09-04; Primary Completion 2015-05-18 (Actual); Study Completion 2015-05-18 (Actual)

PRIMARY OUTCOMES:
Patients with CD will show an increase in the amygdala response to fearful expressions such that the difference between BOLD response in patients and TDs is reduced on MPH relative to placebo. ICU score will be a significant covariate of the inc... | 2 years from the initiation of the protocol
Patients with CD will show an increase in reward prediction errors and reward expected value signaling within striatum and ventromedial frontal cortex (vmPFC) such that the difference between BOLD response in patients and TDs is reduced on MPH r... | 2 years from the initiation of the protocol
Patients with CD will show an increase in conflict related signaling within dorsomedial, lateral and parietal cortices such that the difference between BOLD response in patients and TDs is reduced on MPH relative to placebo. Current ADHD sympto... | 2 years from the initiation of the protocol

SECONDARY OUTCOMES:
Symptom profiles measured by the clinical scales listed in the protocol (CBCL, the ICU, Connor s parent report on ADHD symptom) will be significantly related to the BOLD signal changes after methylphenidate administration. | 2 years from the initiation of the protocol

CONTACTS AND LOCATIONS:
Overall Officials: James J Blair, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)

REFERENCES:
- [Background] Waschbusch DA, Carrey NJ, Willoughby MT, King S, Andrade BF. Effects of methylphenidate and behavior modification on the social and academic behavior of children with disruptive behavior disorders: the moderating role of callous/unemotional traits. J Clin Child Adolesc Psychol. 2007 Oct-Dec;36(4):629-44. doi: 10.1080/15374410701662766. PMID 18088220
- [Background] Blair RJ. Neurocognitive models of aggression, the antisocial personality disorders, and psychopathy. J Neurol Neurosurg Psychiatry. 2001 Dec;71(6):727-31. doi: 10.1136/jnnp.71.6.727. PMID 11723191
- [Background] White SF, Pope K, Sinclair S, Fowler KA, Brislin SJ, Williams WC, Pine DS, Blair RJ. Disrupted expected value and prediction error signaling in youths with disruptive behavior disorders during a passive avoidance task. Am J Psychiatry. 2013 Mar;170(3):315-23. doi: 10.1176/appi.ajp.2012.12060840. PMID 23450288